CLINICAL TRIAL: NCT05413278
Title: Fit for Transfer: Targeted Interventions for Successful Transition and Transfer of Adolescents With Inborn Errors of Metabolism to Adult Metabolic Services
Brief Title: Targeted Interventions for Successful Transition and Transfer of Adolescents With Inborn Errors of Metabolism to Adult Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Fit_for_transfer
Record Dates: First submitted 2022-05-25; First posted 2022-06-10 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Transition; Inborn Errors of Metabolism
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Other): Patient education, empowerment, and information
  Interventions: Behavioral: Behavioral

INTERVENTIONS:
Behavioral: Behavioral — Patient education, information and empowerment

SUMMARY:
Main aims of this project are

* To assess the baseline status-quo of transition and "fitness for transfer" in terms of information about the adult centre and team, organisational and practical skills (blood sampling and sending, how to make an appointment etc.), disease- and treatment-related knowledge, health-related quality of life (HrQoL), and self-efficacy in adolescnets with inborn errors of metabolism. Biochemical or physical parameters as appropriate for the respective diseases from 12 months before are documented.
* To provide targeted, structured intervention modules (using available and, if necessary, adapted materials).
* To measure the effects of these interventions on information about adult services short-term (within a month) and to re-assess all other baseline status-quo parameters long-term (6 and 12 months later). Psychological assessments will be complemented by biochemical or physical parameters as appropriate for the respective diseases and indicative for transition success.

ELIGIBILITY:
Inclusion Criteria:Patients

* with an inborn error of metabolism in the care of a specialized metabolic care unit
* requiring specialized adult metabolic care
* at least 14 years old
* with a disease for which at least one biochemical and / or physical parameter disease marker is well established .

Exclusion Criteria:

Patients -

* with insufficient knowledge of the German
* with cognitive impairment to a degree that consent, and participation would be impossible
* in an end-of-life situation
* with a disease for which no biochemical and / or physical parameter disease marker is well established

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease knowledge | change from baseline to 1 month
  interview, semistructured

CONTACTS AND LOCATIONS:
Locations (8):
- Austria (2):
  - University Childrens Hospital Vienna, Vienna
  - University Hospital Vienna, Vienna
- Switzerland (6):
  - University Childrens Hospital Basel, Basel
  - University Hospital Basel, Basel
  - University Childrens Hospital Bern, Bern
  - University Hospial Bern, Bern
  - University Childrens Hospital Zürich, Zurich
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No